CLINICAL TRIAL: NCT01934530
Title: Implant Associated Soft Tissue Defects in the Anterior Maxilla: A Randomized Control Trial Between Subepithelial Connective Tissue Graft and Acellular Dermal Matrix Allograft
Brief Title: A Randomized Control Trial Testing Connective Tissue Grafts vs. Allograft on Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UM-Anderson-10
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Dental Implant Soft Tissue Defects in the Anterior Maxilla
Keywords: implant complications; esthetics; soft tissue grafting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connective Tissue Graft - Control (Active Comparator): The donor tissue was harvested from tissue palatal to maxillary premolars and anterior to the mesial of the first molars. A horizontal incision corresponding to the width of the recipient bed plus 4mm was made 3 mm apical to the gingival margin. A small secondary vertical incision was tolerated on the mesial aspect of the surgical site to allow for a split thickness technique. The flap was then positioned over the graft and sutured with attempts to cover the grafted tissue to 2mm coronal to the implant/abutment interface pending flap tension. Follow up was monitored over 6 months at various time-points.
  Interventions: Procedure: Soft Tissue Grafting
- Alloderm - Test (Experimental): ADM graft was prepared according to the manufacturer's instructions. The preparation requires rehydration in 50ml sterile saline or Ringers Solution for five minutes and repeated twice. The graft was then transferred to the recipient bed with the basement membrane side facing up and connective tissue on the periosteum. The allograft was trimmed to cover the defect dimensions up to the implant-abutment interface. There was a 4mm margin added to the width on each side to account for lateral contraction as with the connective tissue. With sterile moist gauze, pressure was applied to the graft for proper adaptation to the wound bed. The graft was sutured with a single sling and the flap with a double sling. Simple interrupted sutures were used to close vertical releases.
  Interventions: Procedure: Soft Tissue Grafting

INTERVENTIONS:
Procedure: Soft Tissue Grafting — All patients were treated with infiltration of local anesthetic with vasoconstrictor if noted tolerable by the medical history. Surgeons were then notified if the patient was randomized to the test or control according to a blinded treatment assignment. In both groups, anesthesia was confirmed at the implant site and the palatal donor site if indicated. The recipient bed was then prepared.
  Vertical incisions were made at the defect at line angles and horizontal incisions connected the two vertical releases intrasulcularly without involving the interdental papilla. The flap was reflected as a full thickness flap maintaining the integrity of the collagen attachment with de-epithelialization of papilla to allow for coronal advancement.

SUMMARY:
This randomized controlled clinical pilot trial compared the efficacy of two soft tissue grafting methods for correcting esthetic discrepancies associated with non-molar implants in the maxilla. Specifically, it was explored whether defects treated with connective tissue grafts (SCTG) differed in their outcomes from defects treated with acellular dermal matrix allografts (ADM).

DETAILED DESCRIPTION:
Thirteen patients who presented with implants displaying recession, thin biotype, concavity defects or a combination thereof associated with single crowned dental implants participated in this randomized control trial. The control group (N=7) received SCTG and the test group (N=6) received ADM, both under coronally positioned flaps. Data were collected before surgery, and 6 weeks, 3 months, and 6 months after the surgery. Outcome measures included soft tissue, hard tissue, and esthetics parameters and psychosocial data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of at least 18 years of age
* Maxillary non-molar implant with failing pink esthetic profile
* Implants with adjacent landmarks (only one can be an implant)
* Healthy implants measured by the lack of peri-implantitis and mucositis
* Good oral hygiene.

Exclusion Criteria:

* Unstable systemic diseases, compromised immune system, or unstable bleeding disorders
* History of radiation or cancer in the oral cavity
* Use of IV bisphosphonate or steroid medication
* Use of tobacco products (>1/2 pack per day)
* Pregnancy
* Mucogingival surgery or implant placement within the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-08; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Recession Correction | 6 Months
  Change in recession was recorded at baseline, 6 weeks, 3 months and 6 months after grafting.

SECONDARY OUTCOMES:
Concavity Correction | 6 Months
  At baseline, 6 weeks, 3 months, and 6 months after grafting, buccal concavities were measured.

OTHER OUTCOMES:
Tissue Thickness | 6 Months
  Tissue thickness was measured with a 25 endodontic file with rubber stopper at baseline, 6 weeks, 3 months and 6 months after grafting.
Implant Esthetics | 6 Months
  Implant esthetics were rated with written survey by both the subject and clinician.
Psychosocial Data | 6 months
  Subjects completed questionnaires regarding their quality of life during the study by written survey.

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS, MS, PhD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States